CLINICAL TRIAL: NCT05857735
Title: Kuwait Heart Foundation Registry of Acute Coronary Events
Acronym: KHF RACE
Status: Completed | Type: Observational
Sponsor: Gulf Heart Association (Other)
Collaborators: Servier (Industry); Sanofi (Industry); Beshara company (Unknown); Kuwait Heart Foundation (Unknown)
Responsible Party: Principal Investigator, Mohammad Zubaid, Professor, Gulf Heart Association
Other Study IDs: KHF1
Record Dates: First submitted 2023-05-02; First posted 2023-05-15 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-03

CONDITIONS: ACS
Keywords: Mortality; Inhospital MACE; 30-day MACE

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- ACS patients: Patients admitted to hospital with diagnosis of ACS.
  Interventions: Other: Observational registry with no intervention.

INTERVENTIONS:
Other: Observational registry with no intervention. — No intervention

SUMMARY:
Acute coronary syndrome (ACS) is the most common presentation of Coronary Artery Disease (CAD). It causes significant morbidity and mortality. The Gulf Registry of Acute Coronary Events (Gulf RACE) was conducted in 2007 and filled a wide gap in our understanding of ACS and its management in Kuwait and the Arabian Gulf region. However, the management of ACS has undergone tremendous advances over the last two decades involving pharmacotherapy and device therapy. Practice guidelines have also changed over the last decade. For example, in 2007, there was no catheterization laboratory in any of the general hospitals in Kuwait, primary percutaneous coronary intervention (PCI) was not being practiced, and the rate of in-hospital cardiac catheterization for all ACS patients was very low at around 10%. Currently, of the eight general hospitals in Kuwait, six have catheterization laboratories and five of the six serve as primary PCI centers. There is no contemporary ACS registry in Kuwait, studying its incidence, management, and influence of current changes in clinical practice on patients' outcomes. This multicentre disease-based, country-wide registry is guided by the American Heart Association policy statement for expanding the applications of existing and future clinical registries and the User's Guide published by the Agency for Health care Research and Quality guidance.

DETAILED DESCRIPTION:
This is a prospective, multicentre, country-wide registry of patients who are admitted to any of the eight general hospitals in Kuwait with a diagnosis of ACS over 6-months or more to include 10,000 patients. ACS diagnosis includes ST-segment elevation myocardial infarction (STEMI), non-ST-segment elevation myocardial infarction (NSTEMI) and unstable angina.

The protocol mandates the following basic points:

1. Enrol all consecutive patients who get admitted to hospital.
2. Patients or their relatives should consent for enrolment in the registry.
3. Follow-up of all patients for 30 days from the admission event.

The Principal Investigator has formed a steering committee and drafted a protocol and case report form (CRF). The steering committee members will meet to finalize the protocol and the CRF. Then an investigators meeting will be held to go over the fine details of the protocol and CRF and to instruct the investigators on how to use the online CRFs.

Data entry will be entered online. Quality Control Surveyors will carry out quality control visits. This will involve the inspection of 5% of the data source (hospital files) of enrolled patients against entered patient data for their accuracy. Centres that are identified to be consistently inaccurate will be warned and might be withdrawn from the registry if necessary. This quality control process will be carried out at 1 month and again at 3 months, from the start of the study. It will later be decided whether other subsequent checks would be required. In addition, the Chief Site Officer (CSO) in each hospital will be required to carry out quality control checks at his/her own hospital. This will involve the random checking of 2 files per week involving checking the online CRF and data source.

The different elements of the form will be filled out prospectively during patient stay in the hospital and subsequently at follow-up. All patients will be followed up for 30 days post ACS.

The registry and data collection will be conducted prospectively with the following objectives:

1. Determine the incidence of ACS in Kuwait.
2. Examine the risk factors and outcomes of patients with ACS in Kuwait. Outcomes include mortality, myocardial infarction (MI), cerebrovascular accident (CVA), bleeding, cardiogenic shock, heart failure and others.
3. Study the influence of modifiable and non-modifiable risk factors on outcomes, e.g., influence of age, diabetes, hypertension.
4. Evaluate current ACS practices in Kuwait by examining degree of physician adherence to guidelines of ACS management.
5. Examine the applicability of Global Registry of Acute Coronary Events (GRACE) risk score to our patient populations.
6. Create "Kuwait acute coronary syndrome risk score" (Kuwait risk score), a risk score that better assesses outcomes in our patient population.
7. Compare the effect of current management of ACS in Kuwait, with our previously published data in 2007 on patients' outcomes.
8. Compare our management and outcomes (primary and secondary endpoints) to published international outcomes.
9. Establish a network of hospitals and investigators who are willing to do research. This network will serve as a nucleus for future country-wide projects.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is admitted to hospital with admission diagnosis of ACS.
2. Patient or a relative consent to enrolment in the registry.

Exclusion Criteria:

1- Refusal or inability to consent for enrolment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are admitted to any of the eight general hospitals in Kuwait with a diagnosis of ACS. The sample size will be 10,000 patients. ACS diagnosis includes ST-segment elevation myocardial infarction (STEMI), non-ST-segment elevation myocardial infarction (NSTEMI) and unstable angina.
Sampling Method: Probability Sample
Enrollment: 10812 (Actual)
Dates: Start 2023-05-15 (Actual); Primary Completion 2024-11-25 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Mortality | through study completion, an average of 6 months
  To measure the adverse outcome of in-hospital mortality in ACS patients in Kuwait.
Major Adverse Cardiac Events (MACE) | through study completion, an average of 6 months
  To measure the in-hospital adverse outcomes like myocardial infarction (MI), cerebrovascular accident (CVA), bleeding, cardiogenic shock, heart failure and others in ACS patients in Kuwait.

SECONDARY OUTCOMES:
Mortality | 30 days from discharge
  To measure the adverse outcome mortality 30 days post discharge in ACS patients in Kuwait.
Major Adverse Cardiac Events (MACE) | 30 days from discharge
  To measure the adverse outcomes like myocardial infarction (MI), cerebrovascular accident (CVA), bleeding, cardiogenic shock, heart failure and others 30 days post discharge in ACS patients in Kuwait.
Rehospitalization | within 30 days from discharge
  To measure the rehospitalization rate within 30 days post discharge in ACS patients in Kuwait.
Revascularization | within 30 days from discharge
  To measure the revascularization rate within 30 days post discharge in ACS patients in Kuwait.
Lipid level control | At 6 months from ACS event
  To measure the state of lipid level control at 6 months from ACS event
Efficacy of lipid lowering agents | At 6 months from ACS event
  To review the types and dosages of lipid lowering agents used.

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad Zubaid, Professor, Principal Investigator — Kuwait University
Locations (1):
- Mubarak Al Kabeer hospital, Kuwait City, Kuwait, Kuwait

IPD SHARING:
Plan to Share IPD: Undecided